CLINICAL TRIAL: NCT03013868
Title: CTCs and Novel Target Bio-marker Analysis for Prediction and Monitoring of Metastasis/Recurrence in Post-surgery Colorectal Cancer Patients Using MiSelect R Rare Cell System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MiCareo Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MiC-SRS-CRC-001
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-05

CONDITIONS: Circulating Tumor Cells, CTC
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the growing public awareness and recent progress in multimodality therapy to the colorectal cancer (CRC), CRC still ranks high on the list of the most common and deadly cancers in Taiwan. The cause of CRC mortality is due mainly to the occurrence of distant metastasis. Several reports suggested that circulating tumor cells (CTCs) highly associated with metastasis suggesting that targeting CTCs may offer an unprecedented opportunity to prevent the development of metastasis. Early detection and characterization of CTCs is therefore important as a potential strategy to monitor the progression of CRC. The current proposal is focused on detecting CTCs from peripheral blood of CRC patients using Miselect R system. We will monitor the amount of CTCs and correlate with CRC progression and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 and less than 90 years of age.
2. Colorectal cancer stage II/III patients who will undergo surgical resection.
3. Subject having agreed to participate in the study and follow the study procedures by providing written informed consent prior entering the study.

Exclusion Criteria:

1. Have other cancer history.
2. Subject being identified with any blood borne infectious disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 Colorectal cancer stage II/III patients who will undergo surgical resection
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan